WALANT Versus Local Anesthesia in Central Venous Catheter Insertion

Unique Protocol Id: B.30.2.ATA.0.01.00/830

Document Date: 01.11.2023

Statistical analyses of the study were performed using the IBM SPSS Statistics for Windows, Version 31.0 (Armonk, NY: IBM Corp) package program. The distributional properties of continuous numerical variables were assessed using visual (histogram and Q–Q plot) and analytical (Shapiro–Wilk test) methods. Comparisons between two independent groups were made for non-normally distributed data using the Mann–Whitney U test, and for normally distributed data using the Independent Samples t-test.

Descriptive statistics for non-normally distributed variables were presented as median, 25%–75% quartiles, and minimum–maximum values, and boxplot plots were used for visual assessment of distribution. Normally distributed data were expressed as mean  $\pm$  standard deviation and 95% confidence intervals; error bar graphs were preferred for visual presentation of these variables.

For group comparisons of categorical variables, the Pearson chi-square test or Fisher's exact test was used, depending on the appropriateness of the data. Categorical data were presented as frequency (n) and percentage (%), and were also visualized with bar graphs. In all statistical analyses, a p value of <0.05 was considered statistically significant.